CLINICAL TRIAL: NCT04437992
Title: Feasibility Study of a New Screening Program for Major Aneuploidies (T21, T18, T13) in the Emilia-Romagna Region (SAPERER)
Acronym: SAPERER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: SAPERER
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Autosomal Aneuploidy
Keywords: aneuploidies, down syndrome, Edwards syndrome, Patau syndrome
MeSH Terms: conditions — Aneuploidy; Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome | interventions — dichlorobis(azomycin)platinum II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: * Pregnant women resident in the Emilia Romagna region who access the combined test at regional counseling centers and hospital prenatal clinics.
  * Women able to understand the information, participate in pre-test counseling and provide informed consent.
  Interventions: Genetic: NIPT

INTERVENTIONS:
Genetic: NIPT — The test, which requires two 10 ml tubes of blood, will be performed simultaneously with the chemical biomarkers of the combined test at 10-12 weeks of gestation

SUMMARY:
The study is promoted by the Emilia Romagna Region which identified in the Bologna AUSL the coordinating center (Unità Operativa Complessa Laboratorio Unico Metropolitano, LUM, Maggiore Hospital). The medical genetics centers, participating in the technical-scientific coordination group of assessment (resolution No. 1894, 4/11/2019), the family counseling centers and the region prenatal hospital clinics are involved as collaborative experimental centers.

Currently, 14,400 combined tests are carried out in the Emilia Romagna Region every year.

As a result offering the new non-invasive NIPT test, it is estimated that the number of participants in the screening program will increase by up to 20,000/year.

The study will collect data on the women who will access the combined test in the first 9 months of the protocol and join the enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women resident in the Emilia Romagna region who access the combined test at regional counseling centers and hospital prenatal clinics.
* Women able to understand the information, participate in pre-test counseling and provide informed consent.

Exclusion Criteria:

* Women under the age of 18 and/or unable to give informed consent
* pregnancies with more than two twins
* certain evidence of initial twinning, with subsequent disappearance of one of the twins (vanishing twin)
* known maternal chromosome mosaicisms present in the mother and involving the chromosomes subject to investigation
* presence of neoplasia in pregnant women
* previous allogeneic transplantation in pregnant women
* immunotherapy, radiotherapy or hemotransfusion performed in the pregnant woman within the previous 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Pregnant women resident in the Emilia Romagna region who access the combined test at regional counseling centers and hospital prenatal clinics.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-04-27 (Estimated); Study Completion 2021-04-27 (Estimated)

PRIMARY OUTCOMES:
NIPT | 9 months
  Establish in which percentage invasive tests (amniocentesis and chorionic villus sampling) would be avoidable by replacing routine screening methods (i.e. combined test) with non-invasive prenatal test (NIPT).

SECONDARY OUTCOMES:
Percentage of NIPT | 9 months
  Establish a percentage of NIPT with inconclusive results
diagnostic performance | 9 months
  Verify the diagnostic performance of the Vanadis NIPT method by verification of sensitivity, specificity, and predictive power in comparison to the combined test currently in use
Detection of Chromosomal Abnormalities | 9 months
  Evaluate the added value of nuchal translucency for the detection of Chromosomal Abnormalities other than T21, T18, T13
TAT (turnaround time) | 9 months
  Evaluate TAT (turnaround time) of the NIPT and operability of the technology adopted by the laboratory
Validate NIPT organizational infrastructure | 9 months
  Validate the organizational infrastructure for the NIPT execution in the area outside of the reference laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Regione Emilia Romagna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No